CLINICAL TRIAL: NCT02963103
Title: A Single-center Pilot Study to Assess the Safety and Efficacy of a Tacrolimus Based Immunosuppressive Regimen in Stable Kidney Transplant Recipients Converted From Cyclosporine Based Immunosuppressive Regimen
Brief Title: A Study to Assess the Safety and Efficacy of a Tacrolimus Based Immunosuppressive Regimen in Stable Kidney Transplant Recipients Converted From Cyclosporine Based Immunosuppressive Regimen
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor decision to terminate the study because subject enrollment was difficult.
Sponsor: Astellas Pharma Korea, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRG-KT-10-01
Record Dates: First submitted 2016-10-06; First posted 2016-11-15 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: Kidney Transplantation
Keywords: Tacrolimus; Kidney transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus group (Experimental): oral
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Oral
  Other Names: Prograf (R)

SUMMARY:
The objective of this study is to observe and evaluate the change in renal function following conversion from cyclosporine-based immunosuppressive regimen to tacrolimus-based one.

ELIGIBILITY:
Inclusion Criteria:

* Patients received a kidney transplant at least 12 months before enrollment.
* Patients whose dosage of previous immunosuppressants has not been changed and remained for at least 4 weeks before enrollment, and blood trough level of cyclosporine is 100 to 200 ng/mL.
* Patients who have the side effects (hypertension, hyperlipidemia, gingival hyperplasia and hypertrichosis/hirsutism) during use of cyclosporine.
* Serum creatinine < 2.3 mg/dl at enrollment
* Female patients of childbearing potential must have a negative serum pregnancy test prior to enrollment, and agreed to use effective contraception during the trial.
* Patients considered clinically stable

Exclusion Criteria:

* Patients who have previously received an organ transplant other than a kidney.
* Patients who have had acute transplant rejection within 12 weeks, or acute transplant rejection requiring antilymphocyte therapy within 24 weeks prior to enrollment.
* Patients newly diagnosed malignant tumors after organ transplant, but the patients treated completely with basal or squamous cell carcinoma of the skin are excepted.
* Patients who have an underlying disease such as focal segmental glomerulosclerosis (FSGS) or type II membranoproliferative glomerulonephritis (Type II MPGN).
* Proteinuria > 2 g/24 hrs.
* Patients who have "Creeping creatinine" (a 20% increase in their creatinine for six months before their enrollment).
* Patients whose Alanine Aminotransferase (ALT) and/or Aspartate Aminotransferase (AST) is twice higher than the normal range in the center.
* Patients who have liver cirrhosis.
* Patients who are pregnant or breastfeeding.
* Patients who had been HIV-positive.
* Patients who have a known allergy to Prograf® or its ingredients, steroids or adjuvants.
* Patients who have an unstable medical condition that may affect the evaluation of the study's objectives.
* Patients who are receiving prohibited concomitant medications or who received those medications within 28 days of their enrollment.
* Patients who are currently participating in another clinical trial or who received the investigational drug in another trial within 28 days of their enrollment.
* Patients who are at the risk of drug abuse or mental disorders or communicate difficulties.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-05; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline in GFR | Baseline and Week 24
  GFR: glomerular filtration rate

SECONDARY OUTCOMES:
Change from baseline in total cholesterol | Baseline and Week 24
Change from baseline in Triglycerides | Baseline and Week 24
Change from baseline in LDL | Baseline and Week 24
  LDL: low density lipoprotein cholesterol
Change from baseline in HDL | Baseline and Week 24
  HDL: high density lipoprotein cholesterol
Change from baseline in the number of antihyperlipidemic drugs | Baseline and Week 24
Change from baseline in blood pressure | Baseline and Week 24
Change from baseline in the number of antihypertensive drugs | Baseline and Week 24
Change from baseline in number of participants who have had hirsutism | Baseline and Week 24
  Investigator's judgment
Change from baseline in number of participants who have had gingival hypertrophy | Baseline and Week 24
  Investigator's judgment
Overall incidence rate of adverse events | up to Week 24
Proportion of participants with patient survival | up to Week 24
Proportion of participants with organ survival | up to Week 24
Acute rejection rate confirmed by biopsy | up to Week 24
Ratio of mean dose of cyclosporine to tacrolimus | up to Week 24

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Korea, Inc.
Locations (1):
- KR00001, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided